CLINICAL TRIAL: NCT01575093
Title: Safety Evaluation of Bowel Cleansing Regimen for PillCam® COLON 2 Capsule Endoscopy
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Medtronic - MITG (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: MA-112
Record Dates: First submitted 2012-03-11; First posted 2012-04-11 (Estimated); Last update posted 2019-07-31 (Actual); Status verified 2012-07

CONDITIONS: Healthy Volunteers
Keywords: Healthy volunteers

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: The preparation regimen — Regimen includes administration of 4 Senna tablets 2 days before the procedure, 2-liters of PEG on the evening before the procedure, 2-liters of PEG on the morning of the procedure, 10mg Metoclopramide, two boosts (6-oz and 3-oz) of SUPREP oral sulfate solution and a 10mg Bisacodyl suppository

SUMMARY:
This study is designed to evaluate the safety of a preparation regimen for PillCam® Colon 2 Capsule Endoscopy.

DETAILED DESCRIPTION:
The preparation regimen used for the PillCam® Colon 2 procedure consists of several colon cleansing materials.

Different combinations of the above regimen were tested and evaluated for safety by monitoring of adverse events in multiple clinical studies, with more than 1000 subjects enrolled to date. No Serious Adverse Events related to the preparation were noted.

In this study, each subject will be required to undergo serum chemistry tests (blood tests) at several time points to evaluate the safety of the regimen.

No capsule ingestion is involved.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is between 50 - 75 years of age.
2. Subject is healthy without any known disease, or any current symptoms of any disease or other abnormal condition.
3. Subject received an explanation about the nature of the study and agrees to provide written informed consent.
4. Subject has normal serum chemistry tests at baseline.

Exclusion Criteria:

1. Subject has any allergy or other known contraindication to the medications used in the study.
2. Subject with history or clinical evidence of renal disease and/or previous clinically significant laboratory abnormalities of renal function parameters.
3. Subject has Type 1 or Type II Diabetes.
4. Subject has any condition which precludes compliance with study instructions.
5. Women who are either pregnant or nursing at the time of screening, or are of child-bearing potential and do not practice medically acceptable methods of contraception.
6. Subject suffers from life threatening conditions.
7. Concurrent participation in another clinical trial using any investigational drug or device.

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2012-03; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
To evaluate the safety of a bowel preparation regimen comprised of Sulfate free Polyethylene glycol electrolyte lavage solution (SF-PEG) plus SUPREP oral sulfate solution as a "booster", in adult subjects. | Latest blood test conducted (i.e. 24 hours after suppository or seven days after procedure)
  Safety will be evaluated by number of Adverse Events and percentage of subjects with clinically siginifcant change in serum chemistry test.

CONTACTS AND LOCATIONS:
Overall Officials: PANKAJ K. KASHYAP, M.D., Principal Investigator — Pinnacle Research Group, LLC
Locations (1):
- Pinnacle Research Group, LLC, Anniston, Alabama, United States

REFERENCES:
- See also: Pinnacle Research Group website — http://www.pinnacletrials.com/